CLINICAL TRIAL: NCT05317533
Title: Prevalence of Distal Radial Artery Occlusion (DRAO) in Patients Undergoing Cardiovascular Catheterization Via Distal Radial Access (DRA)
Brief Title: Prevalence of Distal Radial Artery Occlusion in Cardiovascular Catheterization Via Distal Radial Access
Status: Completed | Type: Observational
Sponsor: Wujin People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CLH20220312
Record Dates: First submitted 2022-03-30; First posted 2022-04-08 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Catheterization; Complications; Distal Radial Artery
Keywords: distal radial artery occlusion;cardiac catheterization

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: cardiac catheterization via distal radial artery — cardiac catheterization via distal radial artery

SUMMARY:
Explore the prevalence of distal radial artery occlusion after cardiac catheterization via distal radial artery and the risk factors

DETAILED DESCRIPTION:
Cardiac catheterization via distal radial artery is prevalent worldwide, which can reduce the prevalence of radial artery occlusion. However, the distal radial artery occlusion has not been detected. This study is designed to explore the prevalence of distal radial artery occlusion in patients undergoing cardiac catheterization via distal radial access at 1 day and 3 months after the procedure, which is explored by ultrasound. In addition, the risk factors of distal radial artery occlusion are also analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Palpable distal radial artery

Exclusion Criteria:

* Age ≥ 90years;
* Height≥ 185cm;
* Cardiogenic shock;
* Refuse to sign the written informed consent.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The subjects consist of patients who present to the cardiac catheterization laboratory for an angiogram or percutaneous intervention for the first time.
Sampling Method: Probability Sample
Enrollment: 805 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-12-18 (Actual); Study Completion 2023-12-18 (Actual)

PRIMARY OUTCOMES:
Prevalence of distal radial artery occlusion | 3 months after procedure
  Prevalence of the distal radial artery occlusion is detected using ultrasound

SECONDARY OUTCOMES:
Prevalence of distal radial artery occlusion | 1 day after procedure
  Prevalence of the distal radial artery occlusion is detected using ultrasound
Thickness of distal radial artery | 3 months after procedure
  Comparison of the thickness of distal radial artery intima using ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Gaojun Cai, MD, Study Chair — Cardiovascular department, Changzhou Wujin People's Hospital
Locations (1):
- Changzhou Wujin People's Hospital, Changzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lin Y, Sun X, Chen R, Liu H, Pang X, Chen J, Dong S. Feasibility and Safety of the Distal Transradial Artery for Coronary Diagnostic or Interventional Catheterization. J Interv Cardiol. 2020 Dec 9;2020:4794838. doi: 10.1155/2020/4794838. eCollection 2020. PMID 33380922
- [Result] Sgueglia GA, Di Giorgio A, Gaspardone A, Babunashvili A. Anatomic Basis and Physiological Rationale of Distal Radial Artery Access for Percutaneous Coronary and Endovascular Procedures. JACC Cardiovasc Interv. 2018 Oct 22;11(20):2113-2119. doi: 10.1016/j.jcin.2018.04.045. PMID 30336816
- [Result] Sattar Y, Talib U, Faisaluddin M, Song D, Lak HM, Laghari A, Khan MZ, Ullah W, Elgendy IY, Balla S, Daggubati R, Kawsara A, Jneid H, Alraies CM, Alam M. Meta-Analysis Comparing Distal Radial Versus Traditional Radial Percutaneous Coronary Intervention or Angiography. Am J Cardiol. 2022 May 1;170:31-39. doi: 10.1016/j.amjcard.2022.01.019. Epub 2022 Mar 2. PMID 35248389
- [Result] Prasad RM, Pandrangi P, Pandrangi G, Yoo H, Salazar AM, Ukponmwan E, Kehdi M, Abela G. Meta-Analysis Comparing Distal Radial Artery Approach Versus Traditional for Coronary Procedures. Am J Cardiol. 2022 Feb 1;164:52-56. doi: 10.1016/j.amjcard.2021.10.034. Epub 2021 Nov 20. PMID 34815063
- [Result] Pacchioni A, Mugnolo A, Sanz Sanchez J, Sgueglia GA, Pesarini G, Bellamoli M, Sacca S, Ribichini F, Reimers B, Gasparini GL. Radial artery occlusion after conventional and distal radial access: Impact of preserved flow and time-to-hemostasis in a propensity-score matching analysis of 1163 patients. Catheter Cardiovasc Interv. 2022 Feb;99(3):827-835. doi: 10.1002/ccd.30005. Epub 2021 Nov 16. PMID 34783423
- [Result] Aminian A, Sgueglia GA, Wiemer M, Gasparini GL, Kefer J, Ruzsa Z, van Leeuwen MAH, Vandeloo B, Ungureanu C, Kedev S, Iglesias JF, Leibundgut G, Ratib K, Bernat I, Barriocanal I, Borovicanin V, Saito S. Distal versus conventional radial access for coronary angiography and intervention: Design and rationale of DISCO RADIAL study. Am Heart J. 2022 Feb;244:19-30. doi: 10.1016/j.ahj.2021.10.180. Epub 2021 Oct 16. PMID 34666014
- [Result] Li F, Shi GW, Yu XL, Song RX, Xiao JQ, Huang HM, Li LM, Zhang LY, Gong C, Cai GJ. Safety and efficacy of coronary angiography and percutaneous coronary intervention via distal transradial artery access in the anatomical snuffbox: a single-centre prospective cohort study using a propensity score method. BMC Cardiovasc Disord. 2022 Mar 2;22(1):74. doi: 10.1186/s12872-022-02518-8. PMID 35236288
- [Result] Shi G, Li F, Zhang L, Gong C, Xue S, Song Y, Cai G. Retrograde Recanalization of Occluded Radial Artery: A Single-Centre Experience and Literature Review. J Endovasc Ther. 2022 Oct;29(5):755-762. doi: 10.1177/15266028211067732. Epub 2022 Jan 10. PMID 35001676